CLINICAL TRIAL: NCT02537223
Title: Phase I Trial of BYL719 in Combination With Concurrent Cisplatin-based Chemoradiotherapy in Patients With Locoregionally Advanced Squamous Cell Carcinoma of Head and Neck (LA-SCCHN)
Brief Title: Phase I Study of BYL719 in Combination With Cisplatin and Radiotherapy in Patients With Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX-001
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Locoregionally Advanced
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Alpelisib; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BYL719, Cisplatin, and Radiation Therapy (Experimental): BYL719, orally, at a starting dose of 200-350 mg, once daily, for 7 weeks. Cisplatin, intravenously, at 100 mg/m2 over 1 hour, every 3 weeks for 3 doses. Radiation therapy, Monday to Friday, for 7 weeks.
  Interventions: Drug: BYL719; Drug: Cisplatin; Radiation: Intensity modulated radiation therapy (IMRT)

INTERVENTIONS:
Drug: BYL719
Drug: Cisplatin
Radiation: Intensity modulated radiation therapy (IMRT)

SUMMARY:
This is a phase 1 study (the first step in testing a new drug or combination, to see how safe the drug and/or combination are) of investigational agent BYL719 in patients with locally advanced head and neck cancer (LA-SCCHN) in combination with standard radiation and chemotherapy (cisplatin).

BYL719 is a new drug that is able to bind (attach to) and block a protein called PI3K-alpha. PI3K-alpha is part of an important pathway called EGFR/PI3K/Akt. A pathway is a series of chemical reactions among proteins in the cells that are involved in the support of normal cellular function. If the pathway is too active, due to changes in those proteins, the pathway can lead to tumor cell growth, survival and invasion. BYL719 has been shown to stop cancers in laboratory and animal studies.

This study is the first time BYL719 will be combined with radiation and chemotherapy.

DETAILED DESCRIPTION:
Participants will be screened for eligibility within 30 days of the intended start of the study treatment. Procedures for research purposes done during screening include archival tumor tissue collection for pharmacodynamic and predictive biomarker research and optional HPV status (if not already known).

Eligible participants will take BYL719, by mouth, once a day, starting one week prior to start of radiation and chemotherapy, for 8 weeks. The starting dose of BYL719 is 200 mg. Participants will be asked to record their doses on a study drug diary. Participants will also receive radiation therapy every day from Monday to Friday for 7 weeks.

Chemotherapy (cisplatin) will be given intravenously on Monday of weeks 1, 4, and 7 (48 hour window during weeks 4 and 7).

While receiving the study treatment, participants will have tests and procedures done once every week for safety purposes.

After the end of the study treatment, participants will be asked to visit the centre every 2 weeks up to week 8 for additional tests and procedures for safety purposes. Between week 8-12 after completing the study treatment, participants will have tumor measurements done to assess efficacy.

Participants will continued to be followed every 3 months up to 1 year, then every 6 months for 2 years (total of 3 years).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with study requirements
* Age >= 18 years
* Life expectancy >6 months
* Previously untreated locally advanced squamous cell carcinoma of the head and neck eligible for cisplatin-based chemoradiation
* Not have received prior anti-neoplastic treatment within 2 years
* Resolved toxicities to Grade 1 or less
* Performance status of 0-1
* Adequate organ function
* Able to swallow and retain oral medication

Exclusion Criteria:

* Enrolled on another intervention clinical trial or in prior study within 30 days.
* Taking drugs with risk of prolonging the QT interval or of causing Torsades de Pointes
* Any condition that could increase the risk to the patient by participating which may include:
* Lung disease or uncontrolled hypertension
* Cardiovascular/vascular/cardiac disease
* Uncontrolled severe infection
* Impaired lung function
* Chronic treatment with corticosteroids/immunosuppressive agents
* Not recovered from previous toxicities
* Systemic therapy within 4 weeks of the start of the study treatment
* Active bacterial, fungal or viral infection
* Significant bleeding disorders
* Uncontrolled medical disorder or active infection
* Dementia or significantly altered mental status
* Diabetes mellitus requiring insulin treatment
* Another malignancy within 2 years of the start of the study treatment
* Received live attenuated vaccines within 1 week of the start of the study treatment
* Receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzymes CYP34A or CYP2C8
* Have impaired gastrointestinal (GI) function or GI disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06-14 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Side Effects | 3 years

SECONDARY OUTCOMES:
Time from date of enrollment to date of relapse disease | 3 years
Number of patients who do not have locoregional relapse of disease | 6 months
Number of patients who do not have locoregional relapse of disease | 12 months
Number of patients who do not have a distant metastatic relapse of disease | 6 months
Number of patients who do not have a distant metastatic relapse of disease | 12 months
Time from date of enrolment to date of death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hansen, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada